CLINICAL TRIAL: NCT00276666
Title: Hyperfractionated Accelerated Radiotherapy (HART) With Chemotherapy (Cisplatin, CCNU, Vincristine) for Metastatic (M1-3) Medulloblastoma
Brief Title: Radiation Therapy and Combination Chemotherapy in Treating Young Patients With Metastatic Medulloblastoma Who Have Undergone Surgery
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Children's Cancer and Leukaemia Group (Other)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000454549; CCLG-CNS-2001-06; EU-20577
Record Dates: First submitted 2006-01-12; First posted 2006-01-13 (Estimated); Last update posted 2013-09-17 (Estimated); Status verified 2009-06

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: untreated childhood medulloblastoma
MeSH Terms: conditions — Central Nervous System Neoplasms | interventions — Cisplatin; Lomustine; Vincristine; Chemotherapy, Adjuvant; Radiotherapy

INTERVENTIONS:
Drug: cisplatin
Drug: lomustine
Drug: vincristine sulfate
Procedure: adjuvant therapy
Radiation: radiation therapy

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x-rays to kill tumor cells. Drugs used in chemotherapy, such as lomustine, vincristine, and cisplatin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving radiation therapy together with combination chemotherapy after surgery may kill any tumor cells that remain.

PURPOSE: This phase II trial is studying giving radiation therapy together with combination chemotherapy to see how well it works in treating young patients with metastatic medulloblastoma who have undergone surgery.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the toxicity of hyperfractionated accelerated radiotherapy (HART) in young patients with metastatic medulloblastoma.
* Determine the toxicity of chemotherapy (vincristine during radiotherapy and 8 courses of lomustine, cisplatin, and vincristine after radiotherapy) in association with HART in these patients.

OUTLINE: This is a multicenter study.

* Radiotherapy and vincristine: Beginning 4-6 weeks after surgery, patients undergo hyperfractionated accelerated radiotherapy (HART) twice a day, 5 days a week, for 5 weeks. Patients also receive vincristine IV once weekly for 8 weeks beginning in week 1*. Approximately 6-8 weeks after completion of radiotherapy, patients proceed to maintenance chemotherapy.

NOTE: *The first 7 patients undergo radiotherapy without receiving vincristine

* Maintenance chemotherapy: Patients receive oral lomustine once on day 1 and cisplatin IV over 6 hours on day 1 and vincristine IV on days 1, 8, and 15. Treatment repeats every 6 weeks for 8 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed periodically for 5 years.

PROJECTED ACCRUAL: A total of 29 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven medulloblastoma

  * The following variants of medulloblastoma are also eligible:

    * Nodular/desmoplastic medulloblastoma
    * Medullomyoblastoma
    * Melanotic medulloblastoma
* Metastatic disease, meeting at least 1 of the following criteria:

  * Unequivocal evidence on pre- or post-operative MR scan of supratentorial (stage M2) metastases and/or spinal metastases (stage M3)
  * Tumor cells seen on cytospin analysis of lumbar cerebral spinal fluid (CSF) (stage M1) performed between 15 days and 21 days after surgery

    * Involvement of CSF pathways by tumor is defined as the unequivocal identification of primitive neuroectodermal cells, either on cytological grounds or with a combination of cytological and immunocytological features (e.g., reactivity for GFAP or a neuronal marker, such as synaptophysin)
* Underwent surgery to remove the tumor no more than 6 weeks ago

PATIENT CHARACTERISTICS:

* Hemoglobin ≥ 10 g/dL
* Absolute neutrophil count ≥ 1,000/mm^3
* Platelet count ≥ 100,000/mm^3
* Neurologically stable (or improving) during the week before starting radiotherapy
* Lansky (1-16 years) or Karnofsky (>16 years) performance status 30-100%
* No active infection
* No prior malignant disease
* Not pregnant or nursing
* No syndrome with recognized potential for increased sensitivity to radiotherapy and/or chromosomal fragility
* Not require anesthesia
* No hearing loss or renal impairment that would make the patient unable to comply with 'Packer' chemotherapy protocol

PRIOR CONCURRENT THERAPY:

* No steroids, if possible, at the start of radiotherapy OR on a stable or reducing dose of steroids during the week before starting radiotherapy
* No prior chemotherapy or radiotherapy
* Dexamethasone should not be used as an anti-emetic unless other therapies fail

Ages: 3 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 29 (Estimated)
Dates: Start 2001-11; Primary Completion 2010-03 (Estimated)

PRIMARY OUTCOMES:
Toxicity

CONTACTS AND LOCATIONS:
Overall Officials: Roger Taylor, MD, Study Chair — Cookridge Hospital; Frank Saran, MD — Royal Marsden NHS Foundation Trust; Barry Pizer, MD — Royal Liverpool Children's Hospital, Alder Hey; David Ellison, MD — Northern Centre for Cancer Treatment at Newcastle General Hospital; Susan V. Picton, MD — Leeds Cancer Centre at St. James's University Hospital
Locations (22):
- Our Lady's Hospital for Sick Children Crumlin, Dublin, Ireland
- United Kingdom (21):
  - Birmingham Children's Hospital, Birmingham, England
  - Institute of Child Health at University of Bristol, Bristol, England
  - Addenbrooke's Hospital, Cambridge, England
  - Cookridge Hospital, Leeds, England
  - Leeds Cancer Centre at St. James's University Hospital, Leeds, England
  - Leicester Royal Infirmary, Leicester, England
  - Royal Liverpool Children's Hospital, Alder Hey, Liverpool, England
  - Royal London Hospital, London, England
  - Great Ormond Street Hospital for Children, London, England
  - Royal Manchester Children's Hospital, Manchester, England
  - Sir James Spence Institute of Child Health at Royal Victoria Infirmary, Newcastle upon Tyne, England
  - Queen's Medical Centre, Nottingham, England
  - Oxford Radcliffe Hospital, Oxford, England
  - Children's Hospital - Sheffield, Sheffield, England
  - Southampton General Hospital, Southampton, England
  - Royal Marsden - Surrey, Sutton, England
  - Royal Belfast Hospital for Sick Children, Belfast, Northern Ireland
  - Royal Aberdeen Children's Hospital, Aberdeen, Scotland
  - Royal Hospital for Sick Children, Edinburgh, Scotland
  - Royal Hospital for Sick Children, Glasgow, Scotland
  - Childrens Hospital for Wales, Cardiff, Wales